CLINICAL TRIAL: NCT06352528
Title: A Phase 1, Multicenter, Open-label, Single-dose Study to Assess the Pharmacokinetics of Repotrectinib in Healthy Participants and Those With Moderate and Severe Hepatic Impairment
Brief Title: A Study to Assess the Drug Levels of Repotrectinib in Healthy Participants and Participants With Moderate and Severe Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA127-1070
Expanded Access: NCT05926232 (Available)
Record Dates: First submitted 2024-04-03; First posted 2024-04-08 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Hepatic Impairment; Healthy Volunteers
Keywords: Hepatic Impairment; Healthy Volunteers; Severe; BMS-986472; Repotrectinib; Liver Diseases; Pharmacokinetics
MeSH Terms: conditions — Lymphoma, Follicular; Liver Diseases | interventions — repotrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Moderate Hepatic Impairment (Experimental)
  Interventions: Drug: Repotrectinib
- Group 2: Severe Hepatic Impairment (Experimental)
  Interventions: Drug: Repotrectinib
- Group 3: Normal Hepatic Function (Experimental)
  Interventions: Drug: Repotrectinib

INTERVENTIONS:
Drug: Repotrectinib — Specified dose on specified days
  Other Names: BMS-986472

SUMMARY:
The purpose of this study is to assess the drug levels of a single oral dose of repotrectinib in participants with moderate and severe HI, and in healthy matched control participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion Criteria for all Participants (Group 1, Group 2, Group 3):.

i) Adult female (as assigned at birth) not of childbearing potential or male (as assigned at birth) of any race or ethnicity.

ii) Must have a body mass index between 18 and 40 kg/m2 (inclusive) and body weight ≥ 50 kg at the time of signing the ICF.

- Inclusion Criteria for Participants with Moderate or Severe Hepatic Impairment (Group 1 and Group 2):.

i) Participants have moderate or severe HI or cirrhosis due to chronic hepatic disease and/or prior alcohol use.

ii) Participants have moderate (Group 1), or severe (Group 2) HI as defined by Child-Pugh score.

- Inclusion Criteria for a Matched Healthy Participant (Group 3):.

i) Participant must be free of any clinically significant disease that would interfere with the study evaluations.

ii) Participant must have liver-related laboratory test results within the respective reference ranges or with clinically insignificant excursions therefrom as agreed by the investigator.

iii) Participant must be in good health as determined by past medical history, physical examination, vital signs, ECG, and clinical laboratory safety tests. Clinical laboratory safety tests (eg, hematology, chemistry, and urinalysis) and 12-lead ECGs must be within normal limits or clinically acceptable as judged by the investigator.

Exclusion Criteria:

- Exclusion Criteria for all Participants (Group 1, Group 2, and Group 3):.

i) Any major surgery within 4 weeks of the study intervention administration.

ii) History of drug abuse within 1 year of study intervention administration.

iii) History of alcohol abuse within 1 year of study intervention administration.

iv) Participants who currently smoke, as well as those who have stopped smoking less than 6 months prior to dosing on Day 1.

- Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Days 1 to 11
Time of maximum observed plasma concentration (Tmax) | Days 1 to 11
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) | Days 1 to 11
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Days 1 to 11

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to 28 days following last dose
Number of participants with Severe Adverse Events (SAEs) | Up to 28 days following last dose
Number of participants with physical examination abnormalities | Up to Day 11
Number of participants with vital sign abnormalities | Up to Day 11
Number of participants with electrocardiogram (ECG) abnormalities | Up to Day 11
Number of participants with clinical safety laboratory test abnormalities | Up to Day 11

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Panax Clinical Research, Miami Lakes, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - The Texas Liver Institute, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com